CLINICAL TRIAL: NCT01053143
Title: Bridging Study on Safety and Immunogenicity of an Intramuscular Inactivated, Split Virion Swine-Origin A/H1N1 Influenza Non-Adjuvanted Vaccine in Healthy Adults in India
Brief Title: Study of Swine-Origin A/H1N1 Influenza Non-Adjuvanted Vaccine in Healthy Adults in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GPF14; UTN: U1111-1111-6149 (Other: WHO)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Pandemic Influenza; Influenza A Virus, H1N1 Subtype
Keywords: Influenza; Pandemic Influenza; Swine-Origin Influenza A/H1N1 Non-adjuvanted Vaccine; Influenza A Virus, H1N1 subtype; Adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants aged 18 years and older at enrollment.
  Interventions: Biological: A/H1N1 pandemic influenza vaccine (non- adjuvanted)

INTERVENTIONS:
Biological: A/H1N1 pandemic influenza vaccine (non- adjuvanted) — 0.5 mL, Intramuscular

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of one dose of A/H1N1 non-adjuvanted pandemic vaccine to support registration of the vaccine in India.

Primary Objective:

* To describe the safety profile (injection site reactions and systemic events) of the vaccine within 21 days following vaccination, and serious adverse events throughout the study in all subjects

Secondary Objectives:

* To describe the immune response to the vaccine 21 days after vaccination by hemagglutination inhibition (HAI) testing in all subjects
* To describe the antibody persistence 6 months after vaccination by HAI testing in all subjects.

DETAILED DESCRIPTION:
Each study participant will receive one dose of the study vaccine on Day 0, provide pre- and post-vaccination blood samples at 21 and 180 days for immunogenicity testing and undergo safety follow-up for 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria :

* 18 years of age and above on the day of inclusion
* Provision of informed consent form signed by the participant. If the participant is illiterate, an independent witness is required to sign the consent form.
* Participant able to attend all scheduled visits and comply with all trial procedures
* For a female, if sexually active, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination, until at least 4 weeks after the last vaccination.

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine during the study period (except 6 months follow up)
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C as reported by the participant / parent or legal representative and/or based on medical history
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator
* Previous participation in a trial investigating a vaccine with the swine-origin A/H1N1 influenza strain
* History of influenza infection in 2009-2010
* Receipt of any allergy shots and/or seasonal allergy medication in the 7-day period prior to enrollment (vaccination), or scheduled to receive any allergy shots and/or seasonal allergy medication in the 7-day period after enrollment (vaccination)
* Known pregnancy, or a positive urine pregnancy
* Currently breastfeeding a child
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures

Temporary contraindication to be resolved before vaccination:

- Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety profile in terms of solicited injection site reactions, systemic events, and serious adverse events after administration of A/H1N1 pandemic influenza vaccine. | 7 days post-vaccination and entire study duration

SECONDARY OUTCOMES:
To provide information concerning the immune response to A/H1N1 pandemic influenza vaccine. | 21 days post-vaccination
To provide information concerning antibody persistence 6 months after vaccination with A/H1N1 pandemic influenza vaccine. | 6 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (3):
- India (3):
  - Chandigarh
  - New Delhi
  - Pune

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com